CLINICAL TRIAL: NCT03887351
Title: Frailty in Community Dwelling Older Adults With Heart Failure
Brief Title: Frailty Heart Failure Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jonathan Afilalo, Director, Geriatric Cardiology Fellowship Program, Associate Professor, McGill University, Jewish General Hospital
Other Study IDs: MP-05-2019-1682
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure; Frail Elderly Syndrome
Keywords: frailty, heart failure, mortality, quality of life
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JGH Cohort: This cohort will not be subjected to any intervention.
- RVH Cohort: This cohort will not be subjected to any intervention.

SUMMARY:
A prospective longitudinal cohort study aimed at measuring frailty and its associated risk factors community dwelling older adults aged 65 years or older.

The geriatric domains evaluated will include: frailty status, hearing impairment, visual impairment, polypharmacy, sarcopenia, malnutrition, cognitive impairment, depression, fatigue, sleep difficulties, and disabilities.

The primary outcome is all-cause mortality at 1-year post enrollment.

DETAILED DESCRIPTION:
The overarching research question is as follows: Is frailty predictive of patient-centered outcomes in older adults with heart failure (HF)? Hypotheses regarding this research question are: 1) Frailty is associated with increased 12-month mortality, 2) Frailty is associated with increased 3-month mortality or unplanned hospitalization, 3) Frailty is associated with lower baseline health-related quality of life (HrQOL), and 4) Frailty is associated with worsening HrQOL at 3 months.

There are three specific study objectives. 1) To compare the ability of various frailty measures to predict all-cause mortality, hospitalizations, and HrQOL in patients attending an outpatient HF clinic. 2) To examine the determinants of longitudinal changes in frailty measures over time. Lastly, 3) To examine the clinical and frailty related determinants of fatigue in older adults

A prospective longitudinal cohort study will be conducted at a specialized heart failure (HF) clinic at the Jewish General Hospital (JGH) and Royal Victoria Hospital (RVH). The study aims to measure frailty and its associated risk factors in community dwelling individuals, aged 65 years or older and who have been diagnosed with HF (preserved or reduced ejection fraction) for at least 3 months. The multi-domain geriatric assessment will include questionnaires administered by interview, physical performance tests, body composition analysis using a bioimpedance machine, review of clinically acquired biochemical and imaging tests, and chart review. The geriatric domains evaluated will include: frailty status, hearing impairment, visual impairment, polypharmacy, sarcopenia, malnutrition, cognitive impairment, depression, fatigue, sleep difficulties, and disabilities. Baseline assessment will approximate to 40 minutes of patient contact time while follow up phone interviews at 3 and 12 months will approximate to 20 minutes. Outcome measures such as all-cause mortality, HrQOL, unplanned hospitalization will be assessed at 3 months and 1-year post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling outpatients
* Aged 65 years or older
* A HF diagnosis with preserved or reduced ejection fraction for at least 3 months
* Agreed to participate and signed an informed consent form

Exclusion Criteria:

* Outpatients with a recent hospital admission within 3 months
* Acutely decompensated HF status at the time of their visit
* Received intravenous (IV) diuretics or IV inotropes within 3 months
* A moribund health status with life expectancy less than 3 months
* Scheduled to undergo a major surgical or percutaneous procedure within 3 months
* Implantation of cardiac resynchronization therapy within the past 3 months or intent to place
* Patients with a history of heart transplant, currently on the transplant list or with an left ventricular device
* Severe neuropsychiatric impairments
* Non -English or French speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population is determined using the inclusion and exclusion criteria. Study population will be Montreal based.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
All cause mortality at 12 months | 12 months
  All cause mortality (cardiac and non- cardiac causes) assessed using in hospital chart reviews.

SECONDARY OUTCOMES:
All cause mortality | 3 months
  All cause mortality (cardiac and non- cardiac causes) assessed using in hospital chart reviews.
Unplanned hospitalization at 3 and 12 months | 3 months and 12 months
  Unplanned hospitalization (In hospital stay for a minimum of 48 hours) assessed using in hospital chart reviews and self-reported hospitalization.
Health related quality of life at 3 and 12 months measured using the Short Form Health Survey questionnaire (SF-36) | 3 months and 12 months
  The sub-scales of the SF-36 include, physical functioning, bodily pain, general health, vitality, social and functioning, mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Afilalo, MD, MSc, Principal Investigator — Jewish General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Somech J, Joshi A, Mancini R, Chetrit J, Michel C, Sheppard R, Nguyen V, Walker M, Giannetti N, Sharma A, Maghakian D, Laforest E, Afilalo J. Comparison of Questionnaire and Performance-Based Physical Frailty Scales to Predict Survival and Health-Related Quality of Life in Patients With Heart Failure. J Am Heart Assoc. 2023 Mar 21;12(6):e026951. doi: 10.1161/JAHA.122.026951. Epub 2023 Mar 9. PMID 36892053